CLINICAL TRIAL: NCT01237704
Title: Dysphagia Rehabilitation for Nasopharyngeal Carcinoma Patients Post Radiotherapy: a Randomised-controlled Trial
Brief Title: Dysphagia Rehabilitation for Nasopharyngeal Carcinoma Patients Post Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Queen Elizabeth Hospital, Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Michael Tong, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRF 475210
Record Dates: First submitted 2010-10-28; First posted 2010-11-10 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Nasopharyngeal Carcinoma; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional rehabilitation (TR) (Active Comparator)
  Interventions: Behavioral: Traditional rehabilitation (TR)
- Transcutaneous electrical stimulation (ES) (Active Comparator)
  Interventions: Behavioral: Transcutaneous electrical stimulation (ES)

INTERVENTIONS:
Behavioral: Traditional rehabilitation (TR) — TR rehabilitation will be scheduled three 45-minute sessions per week for 4 weeks with a total of 12 sessions that include Mendelsohn manoeuvre, Shaker's exercise, Effortful swallow and Masako manoeuvre.
  Arms: Traditional rehabilitation (TR)
Behavioral: Transcutaneous electrical stimulation (ES) — Subjects will receive three 45-minute sessions per week for 4 weeks with a total of 12 sessions.
  Arms: Transcutaneous electrical stimulation (ES)

SUMMARY:
In Hong Kong, every 30 and 12.9 in 100,000 males and females respectively has nasopharyngeal carcinoma (NPC). With early detection and advances in medical care, the number of NPC survivors post radiotherapy is rapidly growing in Hong Kong. One of the most distressing consequences post radiotherapy for NPC patients is swallowing disorder, or dysphagia. Dysphagia in NPC patients almost certainly cause frequent chest infection, dehydration, malnutrition and limitations to concurrent treatment such as oral medication. Given the existing large costs NPC patients incur to the healthcare system, dysphagia only serves to further inflate the soaring costs.

In an attempt to reduce dysphagia related costs to the healthcare system, swallowing rehabilitation is offered to NPC patients. Currently, two major swallowing rehabilitation approaches are commonly adopted. The first is traditional rehabilitation, which involves patients performing various oropharyngeal exercises aimed at improving swallowing physiology. The other swallowing rehabilitation approach is transcutaneous electrical stimulation, which entails using small amount of electric current to increase muscle strength while patients are engaged in swallowing activities. These two methods are proven as effective in patients with stroke and head and neck carcinoma patients. Neither of these methods, nevertheless, yields any efficacy studies in treating NPC patients. Yet, clinicians continue to use either one or both rehabilitation methods as swallowing rehabilitation.

This study aims to address the gap in efficacy studies on swallowing rehabilitation for NPC patients post radiotherapy. The research results should provide justification for rehabilitation time, clinicians' efforts, costs involved and resources used in rehabilitating the swallowing difficulties of the NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* able 18 years of age
* undergone primary radiotherapy or chemoradiotherapy as the treatment
* are expected to complete the 12 month follow-up

Exclusion Criteria:

* prior history of head and neck surgery except biopsies of the NP or the neck nodes
* previous history or having a concurrent neoplasm other than NPC
* other severe medical problems that might contribute to dysphagia, e.g. cerebral vascular accident, neuromuscular diseases, respiratory diseases that may cause dysphagia
* present contraindications for the use of electrical stimulation which include pregnancy, pacemaker, other implanted electrodes or significant reflux
* non-oral feeding is contemplated in prior to treatment
* inability to complete the assessment including cognitive impairment
* of a low life expectancy related to NPC or other illnesses
* history of dysphagia prior to radiotherapy or chemoradiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | Up to 1 year after rehabilitation program
  Each subject will undergo Fiberoptic Endoscopic Evaluation of Swallowing (FEES) to identify penetration and aspiration risks of each consistency. Subjects will be assessed on five different consistencies: thin fluids, honey-thick fluids, pureed diet, soft diet and biscuits. Therefore, five penetration-aspiration scores will be generated for each assessment.
  Scores will be obtained at baseline, post rehabilitation, six months after baseline and one year after baseline for comparison.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy - Nasopharyngeal (FACT-NP) | Up to 1 year after rehabilitation program
  The validated FACT-NP is a Chinese QOL questionnaire that evaluates the rehabilitation outcomes specifically for NPC patients. Among the sixteen NPC sub-scale items, seven are specific to dysphagia. The total score and dysphagia specific scores will be analysed.
  Scores will be obtained at baseline, post rehabilitation, six months after baseline and one year after baseline for comparison.
Self-rated Swallowing Score | up to 1 year after rehabilitation program
  A questionnaire based on patient's perception of existing feeding difficulties. Scores will be obtained at baseline, post rehabilitation, six months after baseline and one year after baseline for comparison.
Voice Handicap Index - 30 | Up to 1 year after rehabilitation program
  This self-assessment scale consists of 30 items that measures the voice-related quality-of-life over three domains: functional, physical, and emotional. Scores will be obtained at baseline, post rehabilitation, six months after baseline and one year after baseline for comparison.
Oral Assessment Guide | Up to 1 year after rehabilitation program
  This 24 point tool comprise of eight categories: swallow, voice, lips, saliva, tongue, gingival, teeth and mucous membrane. Each category is rated by a scale of 1 (normal), 2 (some abnormality) and 3 (severely abnormal). Scores can be obtained at baseline, post rehabilitation, six months after baseline and one year after baseline for comparison.
Perceptual Evaluation of Voice | Up to 1 year after rehabilitation program
  Four vocal parameters, overall severity, roughness, breathiness and strain, will be rated on a 10-point equal-appearing interval scale by the attending speech therapists. Scores will be obtained at all 4 assessment time point for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tong, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Elizabeth Hospital, Kowloon